CLINICAL TRIAL: NCT06825832
Title: Efficiency of High Power Laser Versus Pulsed Electromagnetic Therapy on Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Elsayed, PRINCIPLE INVESTIGATOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: laser + electromagnetic field
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Hemiplegic Shoulder Pain; Laser Therapy; Pulsed Electromagnetic Therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- INTERVENTION 1 LASER (Active Comparator): The MLS® Laser Therapy device used in this study is M6 (ASA srl -Arcugnano, Italy), equipped with both a robotized multidiode head (up to 3,3W), able to perform automatic scanning treatments, and an MLS® handpiece (up to 1,1W), aimed to perform manual point to point or scanning treatments. Each treatment includes two stages: the scanning of the frontal and dorsal shoulder area of 93 cm2 each with a robotized multidiode head and a point-by-point process with the manual handpiece with 7 points of 3,14 cm2 area. 3 sessions per week for 4 weeks
  Interventions: Device: high power laser therapy
- INTERVENTION 2 PEMFT (Active Comparator): the PEMF application, with application of low intensity and frequency pulsed electromagnetic fields (PEMF), the portable device PMT QS (ASA Srl, Arcugnano) is used, equipped with Flexa applicators (36 x 21 x 2 cm (L x P x H) - 1.2 kg), programmable frequency from 0.5 to 100 Hz and variable magnetic field intensity from 5% to 100% (from ~2.5 to ~40 Gauss)), two solenoid applicators are placed at the anterior and posterior positions in the patient's shoulders and applied for 25 min at 25 G intensity at a frequency of 50 Hz.3 sessions per week for 4 weeks
  Interventions: Device: pulsed electromagnetic field therapy
- INTERVENTION 3 EXERCISE (Active Comparator): The conventional exercise program for hemiplegic shoulder pain (HSP) is stretching exercise therapy, joint stabilization exercise therapy.3 sessions per week for 4 weeks
  Interventions: Other: Exercise

INTERVENTIONS:
Device: high power laser therapy — The MLS® Laser Therapy device used in this study is M6 (ASA srl -Arcugnano, Italy), equipped with both a robotized multidiode head (up to 3,3W), able to perform automatic scanning treatments, and an MLS® handpiece (up to 1,1W), aimed to perform manual point to point or scanning treatments. Each treatment includes two stages: the scanning of the frontal and dorsal shoulder area of 93 cm2 each with a robotized multidiode head and a point-by-point process with the manual handpiece with 7 points of 3,14 cm2 area.
  Arms: INTERVENTION 1 LASER
Device: pulsed electromagnetic field therapy — the PEMF application, with application of low intensity and frequency pulsed electromagnetic fields (PEMF), the portable device PMT QS (ASA Srl, Arcugnano) is used, equipped with Flexa applicators (36 x 21 x 2 cm (L x P x H) - 1.2 kg), programmable frequency from 0.5 to 100 Hz and variable magnetic field intensity from 5% to 100% (from ~2.5 to ~40 Gauss)), two solenoid applicators are placed at the anterior and posterior positions in the patient's shoulders and applied for 25 min at 25 G intensity at a frequency of 50 Hz.
  Arms: INTERVENTION 2 PEMFT
Other: Exercise — The conventional exercise program for hemiplegic shoulder pain (HSP) is stretching exercise therapy, joint stabilization exercise therapy.
  Arms: INTERVENTION 3 EXERCISE

SUMMARY:
This study will be conducted to determine the effectiveness of high-power laser and pulsed electromagnetic field on hemiplegic shoulder pain

DETAILED DESCRIPTION:
One common problem that often manifests two weeks to two months following a stroke is shoulder pain. It adversely impacts patients' quality of life and hinders their ability to regain motor and sensory function. Psychological alterations and sleep problems, such as depression, anxiety, hypervigilance, fear avoidance, pain catastrophizing, trouble falling asleep, and early awakening, can also occure.

The majority of HSP develop in the first 2 weeks up to 6 months and about 65% of those will continue to experience the problem several months after that .

The actual cause of HSP is uncertain and frequently complex. So far, numerous pathogenic processes have been found that are likely to be associated to HSP: Joint subluxation, adhesive capsulitis, complex regional pain syndrome, rotator cuff injury, spasticity, and other conditions .

In the last few decades, an enormous number of treatment options have been developed due to the multiple etiology of HSP, But there is still a great deal of uncertainty regarding their efficacy because several etiologies probably lead to the same problem .

High power laser therapy is one suggested therapeutic option for shoulder pain HPLT has long been used to treat conditions that low power laser therapy (LPLT) cannot, such as increased microcirculation, accelerated tissue regeneration, decreased swelling, inflammation, and pain, because of its photomechanical, thermal, electrical and bio stimulating effects on deep tissues. Benefits of HPLT over LPLT include higher power, deeper tissue penetration, shorter emission durations, and longer rest intervals that avoid heat buildup.

It is hypothesized that compared to single-wavelength low-level laser therapy (LLLT), Multiwave Locked System (MLS) allows for better penetration and therapeutic efficacy .

Magnetic field therapy enhances local cellular activity, organizes collagen fibers, enhances oxygen use in tissues, and speeds up circulation by enhancing blood vessel vasodilation without raising local temperatures but There is insufficient evidence supporting its efficacy and superiority to physical therapy agents .

To our knowledge this is the first study to determine the efficiency of high-power laser and pulsed electromagnetic field on hemiplegic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

1. HSP patients aged 40-65 years.
2. unilateral hemiplegia for the first time.
3. duration of stroke of more than 6 months.
4. Visual Analogue Scale (VAS) of more than 4.
5. patients with 1-3 degrees of spasticity according to Modified Ashworth Scale (MAS).

Exclusion Criteria:

1. Patients with a history of inflammation-related rheumatic disease
2. cervical radiculopathy
3. cardiovascular disease or cardiac pacemakers
4. uncontrolled siezures or sever arrthymia
5. shoulder operations, or shoulder injection during the previous three months were excluded.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
shoulder range of motion | 4 weeks
  BY DIGITAL GONIOMETER
shoulder pain by visual analogue scale (VAS) | 4 weeks
  It will be used to measure pain intensity for each participant in 3 groups (A, B and C). The VAS is usually presented as a 10 cm horizontal line on which the participants' pain intensity is represented by a point between the extremes of "no pain at all "and "worst pain imaginable . zero means no pain ,ten means worst pain.
shoulder pain and disability | 4 weeks
  by Shoulder Pain and Disability Index (SPADI)

CONTACTS AND LOCATIONS:
Overall Officials: Eman Samir Fayez, PHD, Study Chair — faculty of physical therapy cairo uni; Ahmed Karmallaah Mohamed, PHD, Study Director — faculty of medicine cairo uni
Locations (1):
- Cairo Uni, Giza, Ad Doqi, Egypt